CLINICAL TRIAL: NCT07304492
Title: An Artificial Intelligence Model for Screening and Diagnosis of Renal Tumors Based on Non-Contrast CT
Brief Title: AI for Renal Tumors Using Non-Contrast CT
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yajia Gu, MD, Director, Head of Radiology, Principal Investigator, Clinical Professor, Fudan University
Other Study IDs: 2509-Exp275
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Renal Neoplasms; Renal Cyst
Keywords: Artificial intelligence; Renal Neoplasms; Renal Cyst; Computer tomography
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn whether the artificial intelligence method can automatically identify and diagnose renal lesions using non-contrast CT or opportunistic screening.

DETAILED DESCRIPTION:
This study first establishes an AI model capable of effectively detecting and diagnosing kidney lesions based on a multicenter retrospective cohort study. Then, the AI model is applied to a large-scale real-world retrospective and prospective population to validate and improve its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent an abdominal CT examination.
2. Patients with renal lesions were managed according to standard clinical pathways, which included follow-up, biopsy, or surgery.
3. Malignant lesions were pathologically confirmed; benign lesions were confirmed by either pathological diagnosis or imaging follow-up.
4. No prior treatment had been received for the renal disease.

Exclusion Criteria:

1. Patients refuse to undergo recommended follow-up, biopsy, or surgery, which precluded definitive diagnosis of the renal lesion.
2. Absence of complete pathological confirmation for lesions suspected to be malignant.
3. Patients have received any form of prior treatment for the renal lesion.
4. Poor image quality that hampered diagnostic evaluation.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent an abdominal CT examination.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Building an intelligent diagnostic system for renal diseases based on CT scans. | 1 year
  To construct an intelligent system for the detection of renal mass lesions and their differentiation into cysts, benign, and malignant neoplasms.

SECONDARY OUTCOMES:
Further develop artificial intelligence model to effectively diagnose pathological types of common renal tumors. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided